CLINICAL TRIAL: NCT06614101
Title: Study Enabling the Collection of Clinical Data Necessary for the Second Phase of Development of the Glycemic Measurement Device by Analysis of Exhaled Air
Acronym: BOYDSENSE DATA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/24/0046
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes
Keywords: Blood sugar measurement; exhaled air
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient with type 2 diabetes or non-diabetic patient treated in the Diabetology departments (Experimental)
  Interventions: Other: Exhaled air analysis

INTERVENTIONS:
Other: Exhaled air analysis — The patient takes two breaths into two different Module In a Box devices (one measurement per device) which will give two measurements of the volatile organic compounds in the exhaled air. No estimate of blood glucose by breath will be displayed: the Module In Boxes will be set to only display the indication valid measurement/invalid measurement.

SUMMARY:
A pilot study carried out by the company ALPHA-MOS in 2017-19 showed that the analysis of volatile organic compounds contained in exhaled air could reliably predict blood glucose levels. Subsequently, the company BOYDSense, a subsidiary of ALPHA-MOS, produced the Module In a Box prototypes of portable, non-invasive volatile organic compounds analyzers that could be equipped with an on-board algorithm estimating blood glucose levels. The Toulouse University Hospital conducted the BOYDSENSE-GM study in 2021-2023, in partnership with BOYDSense, aiming to develop the first algorithm for calculating blood glucose levels based on the analysis of the breath of 100 patients living with type 2 diabetes and to carry out a first performance test of the Module In a Box prototype in 30 additional subjects with type 2 diabetes. These recent results confirmed the potential of this innovative blood glucose measurement technology and gave the first indications about the next developments needed to improve its performances. The characteristics of the air exhaled by a human are impossible to simulate. Therefore, further development of the glucose calculation algorithm requires the production of additional clinical data, supporting the carrying out of the present study.

DETAILED DESCRIPTION:
The BOYDSense-DATA+ study consists of measuring the concentrations of volatile organic compounds at the same time as capillary blood glucose measurements carried out as part of routine care of patients with type 2 diabetes and non-diabetic individuals at risk of type 2 diabetes. The volatile organic compounds measurements will be done using the Module In a Box prototypes previously used in the BOYDSENSE-GM study. The reference blood glucose levels will be capillary blood glucose values, measured with a properly calibrated blood glucose meter validated for hospital use.

ELIGIBILITY:
Inclusion Criteria:

* Patient living with type 2 diabete or non-diabetic individuals characterized by overweight/obesity (Body Mass Index >= 25Kg/m²) , admitted in the two departments of the Toulouse University Hospital (Diabetology, Metabolic Diseases and Nutrition as well as Endocrinology, Metabolic Diseases and Nutrition).
* Aged 18 years or more.
* Ability to sign informed consent.
* Affiliation to a social security scheme.

Exclusion Criteria:

* Ongoing respiratory infection.
* Pregnancy or breastfeeding.
* Patient under guardianship, curatorship or safeguard of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Measurements of volatile organic compounds | 19 months
  Measurements of volatile organic compounds in participants' breath, measured by the Module In Box device.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Gourdy, MD, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - Fontaine Salée Hospital, Salies-du-Salat, France
  - Rangueil Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No